CLINICAL TRIAL: NCT03942757
Title: BiLirubin Decrease Under Phototherapy Exposure in the Preterm Newborn in Incubator
Acronym: BLUE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0021
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Preterm Infant; Jaundice, Neonatal; Phototherapy
Keywords: preterm infant; jaundice; bilirubin; phototherapy; educational program
MeSH Terms: conditions — Premature Birth; Jaundice, Neonatal; Jaundice | interventions — Phototherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation before educational program: 100 preterm infant medical records will be studied in a first part of this observational study
  Interventions: Other: bilirubin serum level determination; Other: Phototherapy
- Observation after educational program: An educational program will be implemented in the unit after this first period. 100 preterm infant will be included in a second part of this observational study.
  Interventions: Other: bilirubin serum level determination; Other: Phototherapy

INTERVENTIONS:
Other: bilirubin serum level determination — bilirubin serum level before and after phototherapy treatment will be measured
Other: Phototherapy — Preterm infant < 35 weeks of gestation with a jaundice requiring phototherapy according to NICE guidelines can be included for the duration of the phototherapy treatment.

SUMMARY:
Phototherapy is routinely used in neonatal intensive care units for the treatment of jaundice. Guidelines focus mainly on bilirubin serum levels to start the phototherapy. Only few data are available about clinical management of phototherapy devices and subsequently the impact on bilirubin serum decrease. Especially there are no strong recommendations about phototherapy duration, irradiance measurements, incubator temperature and humidity settings. Various factors can influence irradiance and thus the preterm infant bilirubin serum decrease. This study aims at evaluating the impact of an educational program on the use and efficacy of phototherapy in a neonatal intensive care unit.

DETAILED DESCRIPTION:
Only few data are available about clinical management of phototherapy devices for the treatment of jaundice in the preterm infant.

This study is a prospective, monocentric, observational study. Preterm infant < 35 weeks of gestation with a jaundice requiring phototherapy according to NICE guidelines can be included for the duration of the phototherapy treatment.

The decrease in bilirubin serum level before and after phototherapy treatment will be measured.

This decrease in bilirubin serum level will be assessed for two consecutive periods before and after an educational program on jaundice management of the preterm infant.

The investigators aim at demonstrating that an educational program could improve phototherapy management and result in a higher decrease in bilirubin serum during treatment of the preterm infant with jaundice.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant less than 35 weeks gestation
* preterm infant hospitalized in the neonatal intensive care unit of CHU Amiens-Picardie
* preterm infant placed in an incubator
* preterm infant with a jaundice requiring treatment according to NICE guidelines
* preterm infant with a no hemolytic disease
* preterm infant with informed written consent from the parents

Exclusion Criteria:

* preterm infant more than 35 weeks of gestation
* preterm infant with hemolytic disease
* preterm infant with Jaundice related to a cholestasis
* Jaundice requiring exchange transfusion

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospective, monocentric, observational study. All the preterm infant with a jaundice requiring a treatment with phototherapy could been screened for eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Change in bilirubin serum level (μmol/L/h) | before and 24 hours after start of phototherapy treatment
  Change in bilirubin serum level (μmol/L/h) = (end bilirubin (μmol/L) - start bilirubin (μmol/L)) / delay between the 2 measurements (h)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No